CLINICAL TRIAL: NCT02686931
Title: The Investigation of Children With Developmental Delay and Children's Rehabilitation Common Case: A Longitudinal Study
Brief Title: The Investigation of Children With Developmental Delay and Children's Rehabilitation Common Case
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 102-0474A3
Record Dates: First submitted 2015-02-25; First posted 2016-02-22 (Estimated); Last update posted 2018-01-18 (Actual); Status verified 2017-11

CONDITIONS: Developmental Disabilities
Keywords: Developmental delayed; Orthopedic disease; Longitudinal study
MeSH Terms: conditions — Developmental Disabilities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Control: Control: Normal developmental children with orthopedic disease
- Experimental: Experimental: Developmental delayed children

SUMMARY:
Children with developmental disabilities and children's rehabilitation common case investigation: Long-term follow-up study.

DETAILED DESCRIPTION:
Three fundamental goals of early rehabilitation for children with DD are: optimizing body function within each child's prognostic potential, preventing the development of secondary conditions that impact life-long health, and promoting children's participation in their lives. Knowledge of these developmental patterns of FPLA may be helpful in understanding, anticipating, and managing the problems of these patients. The investigators hypothesize that the course of developmental patterns in Function and Participation in Life Activities (FPLA) of patients with DD evolves with their age. The levels of functional recovery included developmental function, activity, participation, and quality of life (QOL). The aim of this study is to investigate the longitudinal outcomes in patients with DD evaluated by developmental function, activity, participation, and QOL. Additionally, the predictors in the initial stage in determining the final developmental patterns in FPLA of these children will be identified.

ELIGIBILITY:
Inclusion Criteria:

1. Children with aged 0-20 years
2. Control group: Children with orthopedic disease, Experimental group: Children with Developmental disabilities

Exclusion Criteria:

1. Low cooperative with follow-up
2. Low cooperative with clinical assessment
3. Low cooperative with questionnaire writing and data collection

Max Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Control and experimental groups
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2013-01; Primary Completion 2018-12 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Change of Comprehensive Developmental Inventory for Infants and Toddlers(CDIIT) | baseline, six months and one year
  Measurement of CDIIT

SECONDARY OUTCOMES:
Change of Chinese Child Developmental Inventory (CCDI) | baseline, six months and one year
  Measurement of CCDI
Change of Bruininks-Oseretsky Test of Motor Proficiency, Second Edition (BOT-II) | baseline, six months and one year
  Measurement of BOT-II
Change of Quality of upper extremity skills test(QUEST) | baseline, six months and one year
  Measurement of QUEST
Change of Peabody Developmental Motor Scales-2nd Edition(PDMS-II) | baseline, six months and one year
  Measurement of PDMS-II
Change of Pediatric Balance Scale(PBS) | baseline, six months and one year
  Measurement of PBS
Change of Gross Motor Function Measure, 66 items,(GMFM-66) | baseline, six months and one year
  Measurement of GMFM-66
Change of Modified Ashworth Scale (MAS) | baseline, six months and one year
  Measurement of MAS
Change of Spinal Alignment and Range of Motion Measure (SAROMM) | baseline, six months and one year
  Measurement of SAROMM

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Ling Chen, PhD, Principal Investigator — Department of Physical Medicine & Rehabilitation, Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No